CLINICAL TRIAL: NCT05389332
Title: Developing and Testing a Mobile Health Intervention to Promote Sun Protection Behaviors and Skin Examination Among Hispanics
Brief Title: A Mobile Health Intervention Among Hispanics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Zhaomeng Niu, Research Associate, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 132206; Pro2022000533 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-05-17; First posted 2022-05-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cancer of Skin
Keywords: Mobile health
MeSH Terms: conditions — Skin Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Aim 1: Interviews with ten to twelve health care providers and community leaders for a 30-60 minute interview via Zoom and recorded.
  Aim 2: We anticipate recruiting four focus groups (2 English, 2 Spanish) with six to eight participants each for a 60-minute audio-recorded focus group. Ten to twelve individual interviews for a 30-60 minute interview via Zoom and recorded.
  Aim 3: A single-arm design: participants will receive WhatsApp messages about skin cancer for three months. The participants will need to complete a survey with the same questions in the pre-survey along with the acceptability and feasibility measures at three-month and six-month follow-ups.
  Aim 4: A pilot RCT comparing two groups: skin cancer and physical activity and nutrition information. Survey at baseline, three-month and six-month follow-ups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile skin cancer intervention (Experimental): Conduct a pilot of the refined intervention among Hispanics to evaluate the preliminary efficacy of the user-centered mobile skin cancer intervention program.
  Interventions: Behavioral: Hispanics Skin Cancer intervention
- Control group: physical activity and nutrition information (Active Comparator): Participants will complete a baseline survey first; and then they will be randomly assigned into either the intervention group or the control group. After the random allocation participants will receive instructions on how to use WhatsApp and then the intervention. The participants will receive WhatsApp messages about skin cancer for three months with optimal frequencies determined by prior aims and complete a post-intervention survey which contains the same questions in the pre-survey. The participants will be contacted at six months after the baseline survey to complete another survey similar to the post-intervention survey.
  Interventions: Behavioral: Control group: physical activity and nutrition for Hispanics

INTERVENTIONS:
Behavioral: Hispanics Skin Cancer intervention — With the insights from the community, the investigators will then develop the mobile intervention targeting Hispanics at risk for skin cancer to promote sun protection and SSE and get feedback to optimize the intervention. After the random allocation participants will receive instructions on how to use WhatsApp and then the intervention. They will receive WhatsApp messages about skin cancer for three months with optimal frequencies determined by prior aims and complete a post-intervention survey which contains the same questions in the pre-survey. The pilot RCT will be conducted around the spring/summer of Year four of the R00 when UVR is generally the highest in the US. The participants will be contacted at six months after the baseline survey to complete another survey similar to the post-intervention survey.
  Arms: Mobile skin cancer intervention
Behavioral: Control group: physical activity and nutrition for Hispanics — Content will be developed from established websites such as CDC's Division of Nutrition, Physical Activity and Obesity. We selected these topics because they are also of concern among Hispanics and provide an unrelated attention control.
  Arms: Control group: physical activity and nutrition information

SUMMARY:
Hypothesis: More than 80% of the participants (n=40) will complete the intervention at three month (intervention completion) and the six month follow-up (retention rate as feasibility). More than 70% of the participants will report high overall study satisfaction (acceptability) with the intervention and study.

This pre-pilot will inform intervention and procedural refinements for the pilot.

Hypothesis: Participants who receive the intervention (n=57) will report more skin cancer-related preventive behaviors (e.g., mean of summed score of sun protection behaviors such as use of sunscreen, etc.) at three month and six month follow-up compared to those in the control condition (n=57, who will receive general information about physical activity and nutrition).

DETAILED DESCRIPTION:
Aim 1: The investigator will conduct individual interviews among key stakeholders such as health care providers and community leaders to plan a mobile skin cancer intervention among Hispanics. Data will be collected from individual interviews (n=10-12) among key stakeholders and triangulated with data from a funded pilot grant (focus groups and surveys with Hispanic community members) to gather information regarding Hispanics perceptions and behaviors related to skin cancer and suggestions for a WhatsApp intervention.

Aim 2: Employing a user-centered approach to develop a WhatsApp intervention to promote skin cancer risk-reduction behaviors among Hispanics and encourage engagement in the intervention. Use an iterative qualitative (focus groups with Hispanics, n=32; individual interviews with key stakeholders e.g., health care providers and community leaders, n=10-12) process to incorporate input from Hispanics and relevant stakeholders to develop a mobile WhatsApp intervention that is theory- and culturally-guided.

Aim 3: The investigators will evaluate the feasibility and acceptability of this mobile intervention in a single-arm pre-, post-test pilot study among at-risk Hispanics.

Aim 4: Refine the intervention and conduct a pilot RCT (n = 114) using this mobile program among Hispanics at risk for skin cancer and assess the preliminary effects of the mobile intervention at 3-month (intervention completion) and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Self-report as Hispanics
* 18 years or older
* No personal history of skin cancer
* Report more than one skin cancer risk factor
* Do not engage in sufficient sun protection behaviors
* Have not conducted a SSE in the past three months
* Own a smartphone and will be willing to use WhatsApp

Exclusion Criteria:

* Currently being treated for melanoma or nonmelanoma skin cancer

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Sun protection behavior by self-report | The change is being assessed at baseline, three month and six month follow-up intervals
  Mean score of use sunscreen with an SPF 30 or higher, seek shade, wear protective clothing, wear wide-brimmed hat, wear sunglasses

SECONDARY OUTCOMES:
Seek shade behavior by self-report | The change is being assessed at baseline, three month and six month follow-up intervals
  Seek shaded areas
Wear protective clothing behavior by self-report | The change is being assessed at baseline, three month and six month follow-up intervals
  Wear protective clothing
Wear wide-brimmed hat behavior by self-report | The change is being assessed at baseline, three month and six month follow-up intervals
  Waer a wide brim hat
Wear sunglasses behavior by self-report | The change is being assessed at baseline, three month and six month follow-up intervals
  Wear sunglasses
Skin self-examination | Changes at baseline, three month and six month follow-up intervals
  Skin examination by oneself
Skin examination by a health care professional | Changes at baseline, three month and six month follow-up intervals
  skin examination by a health care professional

CONTACTS AND LOCATIONS:
Overall Officials: Zhaomeng Niu, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No